CLINICAL TRIAL: NCT05545878
Title: Evaluation of the Effectiveness of the Super Enhanced Single Vision Lens L01 (SESL01) in Reducing Symptoms of Computer Vision Syndrome (CVS): a Double-blind Two-arm Parallel Randomised Controlled Trial
Brief Title: Impact of 'SESL01' Lens on Computer Vision Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Rupal Lovell-Patel, Principal Investigator, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Health 0360
Record Dates: First submitted 2022-09-09; First posted 2022-09-19 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Computer Vision Syndrome
Keywords: Enhanced; Single; Vision; Spectacle; Lenses
MeSH Terms: interventions — Eyeglasses

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomised controlled trial. Participants will be required to have a full eye exam at the UCLan Eye Health Clinic to assess eligibility to enrol in the study. Once participants have been screened and completed the Computer Vision Syndrome Questionnaire (CVS-Q), ensuring that they meet the inclusion criteria, they will be randomly allocated to the Intervention or Control Groups. After the eye exam and CVS-Q score, eligible participants will have the following tests measured as baseline data:1. LogMAR Vision and Visual Acuity (6/6 minimum monocular distance VA and N6 monocular). 2. Monocular and binocular amplitude of accommodation. 3. Near point of convergence. 4. Wilkins Rate of Reading. 5. Accommodative Facility in cycles per minute. 6. Thomson Clinical Eye Tracking. The tests and CVS-Q will be repeated at intervals of 4 weeks for a further three times. The 4-week interval period will start from the date of the spectacle collection.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The procedure adopted in this study for assuring the allocation concealment will be the use of sequentially numbered, opaque, and sealed envelopes (SNOSE).
  Blinding : In our study, the clinicians (opticians) performing the assessment and follow-up and the patients receiving and wearing the spectacles will be blinded to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Super enhanced single vision lens 01 for spectacles (Experimental): Participants in the intervention group will wear the newly designed SESL01 lens with anti-reflection coating. Participants will be asked to wear their spectacles for all daily tasks as normal including when looking at digital screens and near tasks.
  Interventions: Device: Super enhanced single vision lens 01 for spectacles
- Control: Standard single vision lenses with an anti-reflection coating (No Intervention): Participants in the control group will be corrected with standard single vision lenses with an anti-reflection coating. Participants will be asked to wear their spectacles for all daily tasks as normal including when looking at digital screens and near tasks.

INTERVENTIONS:
Device: Super enhanced single vision lens 01 for spectacles — This is a spectacle lens designed to have a small amount of positive power towards the bottom of the lens as this is the area that is in line with the eye when downwards for near tasks such as looking at a digital device.
  Arms: Intervention: Super enhanced single vision lens 01 for spectacles

SUMMARY:
The increased use of digital devices such as computers, smart-phones, tablets, and laptops has transformed how people learn and work and has increased the use of screens. This has created visual challenges for some users, such as maintaining a clear vision for a long period even when looking at different devices. Consequently, digital device users can experience eye problems such as blurred vision, eye strain, headaches, and dry eyes. Such problems are more common in people aged 21-45, and it seems that the COVID-19 pandemic has worsened them.

Studies suggest that using specially designed lenses could reduce these problems. Therefore, the investigators aim to study whether specially designed lenses are more effective than standard ones in minimising these problems. The study will be conducted at the University of Central Lancashire at the Preston campus (UK). The study will recruit 300 participants, divided into two equal groups. Participants in group A will receive spectacles with special lenses while group B will receive spectacles with standard lenses. All Participants will be assessed three times, at 4-week intervals, and the final analysis will be performed at 14 weeks. The reduction of the eye problems will be assessed using a validated questionnaire which will produce a score that will be compared between the two groups at the end of the study.

The study's potential benefits are twofold:

1. Patients using the new lenses will hopefully see a reduction in eye problems
2. Opticians will provide be able to provide better patient care.

DETAILED DESCRIPTION:
Background What is the problem to be addressed? In the last two decades, the way people acquire information has changed dramatically. During that time, engagement with digital devices in developed countries has increased significantly, particularly in the field of mobile media. The increasing use of digital devices showed implications for health, eyes, and vision. A European study found out that by the age of 3, 68% of children regularly use a computer and 54% undertake online activities. In 2016, it was estimated that UK adults typically spend almost 5 hours a day using digital media, with a similar pattern developing in the USA.

The use of digital devices has caused Computer Vision Syndrome (CVS), also called Digital Eye Strain (DES) or Visual Fatigue (VF), which has been well described in the literature for over 20 years.

What is Computer Vision Syndrome? The American Optometric Association defines Computer Vision Syndrome (CVS) as a group of eye and vision-related problems resulting from prolonged exposure to digital/computer devices. CVS has been linked to using a variety of digital devices such as computer/laptop screens, tablets, and smart-phones, which has been steadily growing. The most common symptoms are eye strain, tired eyes, irritation, burning sensation, redness, blurred vision, and double vision. Therefore, a person using digital devices and complaining about one or more of those symptoms might be suffering from CVS. Furthermore, CVS could cause non-ocular symptoms such as headaches and pain in the shoulders, neck, and/or back. Research has identified four CVS categories. The first is asthenopia: eye strain, tired eyes, and dry eyes. The second is ocular and related to eye surface: watery eyes, irritated eyes, contact lens problems. The third is the visual category: blurred vision and slowness of focus. The fourth category is extraocular and is represented by neck, shoulder, and back pain.

CVS symptoms result in poorer visual performance, and even though they are transient, they occur frequently and cause considerable discomfort for sufferers. CVS lowers productivity (increased errors and more frequent breaks) and impinges on job satisfaction and quality of life. Millions of individuals of all ages are at risk of CVS, and according to different studies, the prevalence of CVS ranges from 25% to 93%, depending on the cohort of the studied population, the definition and methodology employed to measure CVS. These results indicate that a large proportion of the population may need treatment for CVS.

CVS affects all age groups, including older age groups (aged 65+), in which the use of technology is also rapidly growing. However, the most affected population are younger users, who are more likely to simultaneously use two or more digital devices. For example, recent US data indicates that while adults aged 60 years and over prefer using laptops and desktop computers, younger adults are more likely to use smart-phones too. Since they use digital devices for work and social purposes (e.g. social media), they often multitask and switch between different devices.

The COVID-19 pandemic introduced homeworking and remote learning and further increased exposure to digital screens. Moreover, lockdown increased unhealthy digital recreational activities, with people turning to television and social media for entertainment.

Management of Computer Vision Syndrome CVS management includes correction of refractive error and/or presbyopia (long-sightedness caused by loss of elasticity of the lens of the eye, occurring typically in middle and old age; managed by prescribing a 'near add'), dry eye management, regular screen breaks, and eye exercises for vergence and accommodative problems (such as a lag in changing the focus from near to far distance). Some studies have explored the role of blue light-filtering spectacle lenses with mixed results, indicating that blue light-filters may not alleviate symptoms of CVS. Given the high prevalence of CVS and near-universal use of digital devices, it is essential that eye care practitioners can provide advice and management options that are evidence based.

Aim To evaluate the effectiveness of the Super Enhanced Single Vision Lens 01 (SESL01) in reducing symptoms of Computer Vision Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* 21-45 years of age
* Adults diagnosed with CVS: CSV-Q score ≥6
* Participants WITH AND WITHOUT refractive error are acceptable BUT none should have previously worn a "near add" correction (e.g. no previous bifocal/varifocal/enhanced single vision lens [ESL] wear)
* Range of refractive errors should be no more than +4.00 to -6.00 dioptric spherical power (DS) and +2.00 dioptric cylindrical power (DC)
* Must use digital devices for work and/or leisure for at least 1 hour per day (this includes smart-phones, tablets, and laptops but EXCLUDES those using desktop computers only)
* Patients MUST have visual symptoms associated with digital device use, e.g. one or more of the following symptoms:

  * Tired eyes
  * Eye strain
  * Blurred vision
  * Frontal headaches
  * Difficulties keeping clear vision when changing focus from near to distance
  * Difficulties keeping clear vision when changing focus from one device to another

Exclusion Criteria:

* Lack of capacity to provide informed consent.
* Amblyopia
* Pregnancy
* Diagnosed dry eye disease

  o If a patient develops dry eye symptoms or is diagnosed at follow-up appointments, treatment will be started and assessed in two weeks.
* On anti-depressants (or other medication that can affect accommodation, such as reduced focusing power)
* Any diagnosed ocular pathology (such as glaucoma, corneal dystrophies, lid disorders, and retinal pathologies)
* Change in ±0.75DS/DC in the spectacle prescription

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Reduction in Computer Vision Syndrome Questionnaire (CVS-Q) score. | 16 weeks
  Is the SESL01 lens effective in reducing the symptoms of the CVS compared with standard single vision lenses, assessed by the reduction in Computer Vision Syndrome Questionnaire (CVS-Q®) scores?
  CVS-Q has 16 ocular and visual related symptoms. The frequency of these symptoms is defined based on how often they occur: sometimes or occasionally, once per week, always or often if they occur two to three times per week or every day. The intensity of the symptoms is scored as never=0, mild to moderate=1, severe=2. To measure the frequency of the symptoms, patients will be asked to choose the following options for each of them: never=0, sometimes or occasionally=1, always or often=2. Participants with a total score of 6-12 were deemed to have mild CVS, those with a score of 13-19 moderate, and those with a score ≥20 were considered to have severe CVS

SECONDARY OUTCOMES:
Is there an increase in accommodative facility value when using digital devices? | 16 weeks
  Is the SESL01 lens effective in improving near visual performance when using digital devices, compared with standard single vision lenses, assessed by clinical measurement of accommodative facility using the standard ± 2.00 dioptre spherical lens flippers, measured as cycles per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Health Clinic, University of Central Lancashire, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.

REFERENCES:
- [Derived] Lovell-Patel R, Ajiboye A, Manfrin A. Evaluation of the effectiveness of the Super Enhanced Single Vision Lens 01 (SESL01) in reducing symptoms of computer vision syndrome (CVS): A study protocol for a double-blind, two-arm parallel randomized controlled trial. Contemp Clin Trials. 2023 Feb;125:107046. doi: 10.1016/j.cct.2022.107046. Epub 2022 Dec 10. PMID 36509248

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT05545878/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT05545878/ICF_001.pdf